CLINICAL TRIAL: NCT03485183
Title: The Effect of White and Pink Noise on Hospitalized Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Callie Rebecca Sullivan, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300001385
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Delirium in Old Age
Keywords: delirium; white noise; pink noise
MeSH Terms: conditions — Delirium | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be recruited for the intervention group and receive the intervention. Their data will be compared to baseline data--data without personal identifiers retrieved from chart review. These data will serve as the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The PI will set up the PicTek white/pink noise machine on the bedside table, and it will automatically turn on at 2200 and off at 0700 to the patient's preferred sound. The staff nurses will chart Nu-DESC scores every shift and as needed for change in mental status as is the current policy. The PI will collect Nu-DESC scores for the duration of the participants' hospital stays, age, race, gender, presence of a dementia diagnosis, and use of a pharmacological sleep aid.
  Interventions: Device: White/Pink Noise
- Control Group (Other): The PI will perform a chart review of patients who were admitted the month prior to the intervention being implemented. The PI will collect Nu-DESC scores for the duration of the participants' hospital stays, age, race, gender, presence of a dementia diagnosis, and use of a pharmacological sleep aid. These patients will receive the standard of care for delirium prevention.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: White/Pink Noise — White and/or pink noise will be played from 2200 to 0700 using the PicTek® white noise machine.
  Arms: Intervention Group
Other: Control Group — Standard of care including lights on during the day and off at night, getting the patient out of bed for meals, presence of a large wall clock in the room, updating the whiteboard with current day, consistent reorientation of patient, geriatrician consults as needed, and pain management.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if using an over-the-counter, commercially available sleep noise machine playing pink or white noise will reduce the incidence of delirium in hospitalized patients over the age of 65. Delirium is an acute change in cognition which commonly occurs in hospitalized older adults, and is linked with sleep-wake cycle disturbance. Delirium is associated with increased morbidity and mortality as well as longer hospital stays. This project will record delirium screening scores for those receiving the intervention and comparing them to baseline data. Reducing delirium rates using a noninvasive, inexpensive method in a hospital setting could have a significant impact on patient outcomes and potentially reduce costs associated with longer hospital stays. It is anticipated that white/pink noise played at night will decrease rates of delirium in hospitalized older adults.

DETAILED DESCRIPTION:
The purpose of this study is to determine if using an over-the-counter, commercially available sleep noise machine playing pink or white noise will reduce the incidence of delirium in hospitalized patients over the age of 65. Delirium is an acute change in cognition which commonly occurs in hospitalized older adults, and is linked with sleep-wake cycle disturbance. Delirium is associated with increased morbidity and mortality as well as longer hospital stays. This project will record Nursing Delirium Screening (Nu-DESC) scores for those receiving the intervention and comparing them to baseline data. Reducing delirium rates using a noninvasive, inexpensive method in a hospital setting could have a significant impact on patient outcomes and potentially reduce costs associated with longer hospital stays.

This protocol is based on two concepts. The first is that white/pink noise aids in promoting both sleep quality and quantity and the second is that poor sleep is associated with delirium. Therefore, it stands to reason that improving sleep may decrease the rate of delirium. It is well documented that the elderly are affected by delirium more than other demographics, therefore the benefits to this group would be the greatest in terms of decreasing morbidity and mortality.

White/pink noise was first described as a successful sleep intervention more than 30 years ago in a cardiac intensive care unit study. From that time to present there have been many studies that describe positive effects on sleep by noise machines as a single intervention, but typically they are bundled with other interventions such as earplugs and eye masks. Within the last 5 years, there has been a resurgence in the clinical study of white/pink noise on sleep quality and many of these studies use the gold standard of polysomnography, which employs many sensors to continuously monitor brain waves and sleep patterns. These studies also show a positive impact on both duration and quality of sleep.

More than 15 recent studies were identified that found a correlation between the sleep cycle and delirium. In these studies, sleep disturbance is present in the majority of patients with delirium. There is a clear link between sleep-wake cycle disturbance and delirium, but it is unclear whether an interrupted sleep-wake cycle causes delirium or vice versa. Despite the uncertainty, studies do show that sleep-enhancing interventions decrease rates of delirium and the duration of the delirium. The principal investigator would like to determine if white/pink noise can improve sleep quality and/or quantity, thereby decreasing the incidence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 65 years of age or older
* have an estimated hospital stay of 3 or more nights
* have no known hearing deficits or wear hearing aids
* be free of delirium on admission
* be legally able to consent

Exclusion Criteria:

* non-English-speaking
* less than 65 years of age
* have known hearing deficits or wear hearing aids
* have delirium on admission
* cannot legally consent to participation
* transferred to/from the ICU before/during being enrolled in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Nursing Delirium Screening Scale (Nu-DESC) Score | Collected every 12-hours shift and as needed for acute change in mental status from baseline through discharge for a minimum of 3 nights not to exceed 14 days.
  Nursing Delirium Screening Scale (Nu-DESC) scores, which are already routinely charted by staff nurses, will be collected after the PI sets up the white/pink noise intervention. A score of >2 is indicative of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Latricia D Weed, PhD, Principal Investigator — Troy University
Locations (1):
- UAB Highlands Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available at this time since this is a small study. The protocol can be made available to other researchers at their request without the inclusion of IPD ensuring participant privacy.